CLINICAL TRIAL: NCT00390494
Title: Outcome From Fibroid Therapies: A Comparison With Normal Controls
Brief Title: Questionnaire Study to Assess Quality of Life After Treatment of Fibroids
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Walter Reed Army Medical Center (U.S. Federal Agency); Georgetown University (Other); The Cleveland Clinic (Other); University of Pittsburgh (Other)
Organization: Walter Reed Army Medical Center (U.S. Federal Agency)
Other Study IDs: 04-44020; A-12818.2a
Record Dates: First submitted 2006-10-17; First posted 2006-10-19 (Estimated); Last update posted 2008-06-30 (Estimated); Status verified 2008-06

CONDITIONS: Leiomyoma
Keywords: Fibroids; Leiomyoma; Hysterectomy; Myomectomy; Uterine Fibroid Embolization; Questionnaire
MeSH Terms: conditions — Leiomyoma | interventions — Hysterectomy; Uterine Myomectomy

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: Hysterectomy
Procedure: Myomectomy
Procedure: Uterine Fibroid Embolization

SUMMARY:
The purpose of this study is to determine the change in symptoms and health-related quality of life in patients undergoing treatment for fibroids. Results from the questionnaire will be compared with results obtained from patients who do not have fibroids in order to determine a score range that differentiates these two groups.

DETAILED DESCRIPTION:
Uterine fibroids are the most common benign uterine tumor affecting approximately 70% of all women in the United States. Sixty percent of the 600,000 hysterectomies performed in the United States annually are done because of uterine fibroids. Hysterectomy has been the definitive treatment for fibroids and has been demonstrated to be effective in controlling symptoms. However, there have been few studies comparing the outcome of hysterectomy to other surgical and non-surgical therapies or to the outcomes experienced by a "normal" population, i.e. those not diagnosed with fibroids. Similarly, the relative effectiveness of myomectomy and uterine fibroid embolization has not been evaluated in the context of other fibroid therapies and minimally invasive variations. Fibroid symptoms experienced by patients are subjective and have not been shown to correlate with fibroid number, size, location, or any other clinical measure of fibroids. As symptoms and their impact are the primary outcomes experienced by patients, a validated questionnaire to measure this impact is needed.

The Uterine Fibroid Symptom and Quality of Life Questionnaire (UFS-QoL) was developed from focus groups of women with leiomyomata. The original items captured key symptoms and areas of life impact voiced by the focus group participants. Content validity was established through cognitive debriefings of women with leiomyomata and review by expert clinicians. The UFS-QoL was then validated in a patient population of women with leiomyomata as well as "normal" controls.

Using the UFS-Qol as the primary measure, this study will provide the basis of comparison for women with uterine fibroids both before and after therapy. "Normal" scores will be established from patients without fibroids. These data will provide the basis for comparing these outcomes to those resulting from a variety of investigational therapies. It will also provide insight into the progression of fibroid-related symptoms in patients established as normal at baseline.

The objectives of this study are:

A. To determine the change in symptoms and health-related quality of life in patients undergoing hysterectomy, myomectomy, and uterine fibroid embolization.

B. To compare the outcomes of each intervention with a normal control group as well as with the other therapies.

C. To validate the UFS-QoL questionnaire in a normal population to determine a normal score range.

D. To validate the UFS-QoL questionnaire in hysterectomy patients to determine a "normal" score for patients without a uterus.

ELIGIBILITY:
Inclusion Criteria: Fibroid Treatment Group

* Pre-menopausal
* Between the ages of 35 and 50, inclusive
* Scheduled to undergo hysterectomy, myomectomy, or uterine fibroid embolization for treatment of uterine fibroids at one of the participating institutions
* Willing to provide written informed consent
* Able to speak and read English

Inclusion Criteria: Normal Control Group (patients not diagnosed with fibroids)

* Pre-menopausal
* Between the ages of 35 and 50, inclusive
* Normal gynecologic examination at time of enrollment with regular menstrual cycle at the time of enrollment
* Willing to provide written informed consent
* Able to read and speak English

Exclusion Criteria: Fibroid Treatment Group

* Currently pregnant
* Cognitive impairment that would interfere with completing the questionnaire
* Severe psychiatric co-morbidity
* Co-morbid or life-threatening condition with life expectancy to be less than 1 year
* Active duty military healthcare beneficiary

Exclusion Criteria: Normal Control Group

* Currently pregnant
* Presence of other gynecologic-related diseases (e.g. endometriosis, pelvic inflammatory disease)
* Cognitive impairment that would interfere with completing the questionnaire
* Severe psychiatric co-morbidity
* Co-morbid or life-threatening condition with life expectancy to be less than 1 year
* Active duty military healthcare beneficiary

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2005-12; Study Completion 2010-12

CONTACTS AND LOCATIONS:
Overall Officials: James B Spies, MD, Study Director — Georgetown University Hospital; LTC G. Larry Maxwell, MD, Principal Investigator — Walter Reed Army Medical Center; Richard Guido, MD, Principal Investigator — University of Pittsburgh; Linda D Bradley, MD, Principal Investigator — The Cleveland Clinic
Locations (4):
- United States (4):
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Magee-Womens Hospital, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Spies JB, Bradley LD, Guido R, Maxwell GL, Levine BA, Coyne K. Outcomes from leiomyoma therapies: comparison with normal controls. Obstet Gynecol. 2010 Sep;116(3):641-652. doi: 10.1097/AOG.0b013e3181ed36b3. PMID 20733447